CLINICAL TRIAL: NCT06212232
Title: Efficacy of a New Piezoelectric Technique in Third Molar Surgery and Evaluation of Postoperative Sequelae: a Randomized Split-mouth
Brief Title: A New Piezoelectric Technique in Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amerigo Giudice (Other)
Responsible Party: Sponsor-Investigator, Amerigo Giudice, Professor, University Magna Graecia
Organization: University Magna Graecia (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 123/2023
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Tooth Diseases; Piezoelectric Technique; Tooth, Impacted; Tooth Extraction Status Nos; Tooth Avulsion; Facial Swelling
Keywords: third molar surgery; facial swelling; 3D facial swelling evaluation; Piezoelectric technique; tooth impacted; piezosurgery
MeSH Terms: conditions — Tooth Diseases; Tooth, Impacted; Tooth Avulsion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Test Group (Experimental): Use of a new piezoelectric technique in third molar surgery
  Interventions: Procedure: Piezoelectric surgery
- Traditional: Control Group (Active Comparator): Use of the traditional technique in third molar surgery
  Interventions: Procedure: Piezoelectric surgery

INTERVENTIONS:
Procedure: Piezoelectric surgery — Application of a new piezoelectric technique in third molar surgery

SUMMARY:
The present study aims to analyze the effect of the piezoelectric technique in third molar surgery in terms of facial swelling, trismus and pain in a split-mouth randomized controlled clinical trial

DETAILED DESCRIPTION:
The present study aims to analyze the effect of of the piezoelectric technique n third molar surgery in terms of facial swelling, trismus and pain in a split-mouth randomized controlled clinical trial. Facial swelling will be assessed using an innovative three-dimensional digital technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 32 years who required both M3M extractions were recruited
* Good health status
* Indication to surgical extraction of both M3M
* Complete root formation
* Surgical risk level classified as "Conventional" or "Moderate" according to - Daugela et al. classification

Exclusion Criteria:

* Person under the age of 18 or over 32
* Allergy or contraindications to administration of corticosteroids
* Acute infection in any of the teeth to be extracted
* Patients with chronic liver disease, diabetes, immune system dysfunction, or haematological disease
* Pregnancy or breastfeeding
* History of treatment with antiresorptive drugs
* Chronic kidney disease

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Facial swelling qualitative analysis | Change from baseline (before surgery) at 2 day after surgery and at 7 days after surgery
  To compare the effectiveness of piezosurgery in reducing facial swelling using qualitative three-dimensional analysis (measured by colorimetric variation given by the overlapping volumes) .
Facial swelling quantitative analysis - volumetric differences | Change from baseline (before surgery) at 2 day after surgery and at 7 days after surgery
  To compare the effectiveness of piezosurgery in reducing facial swelling using quantitative three-dimensional analysis ( volumes measured in cm3) .
Facial swelling quantitative analysis - linear differences | Change from baseline (before surgery) at 2 day after surgery and at 7 days after surgery
  To compare the effectiveness of piezosurgery in reducing facial swelling using quantitative three-dimensional analysis (linear differences measured in cm2) .

SECONDARY OUTCOMES:
Trismus analysis | Change from baseline (before surgery) at 2 day after surgery and at 7 days after surgery
  To assess the effects of piezosurgery on trismus (measured in cm)
Pain analysis with Visual analogue scale (VAS) | Change from baseline (before surgery) at 2 day after surgery and at 7 days after surgery
  To assess the effects of piezosurgery on pain (measured by VAS-score from 0 to 10 point, with 10 as the worst outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Magna Graecia University of Catanzaro, Catanzaro, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: No